CLINICAL TRIAL: NCT03551613
Title: Effect of Honey Supplementation on Serum Leptin in Malnourished Infants and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, yasmin gamal el gendy, Lecturer of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6879990
Record Dates: First submitted 2018-03-19; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Malnourished Infants and Childern

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- honey group (Active Comparator): malnourished children supplemented with honey in dose of 2ml/kg
  Interventions: Dietary Supplement: honey supplementation
- malnourished control group (Placebo Comparator): no honey supplementation only nutrition rehabilitation
  Interventions: Dietary Supplement: honey supplementation
- healthy children (No Intervention): healthy children with no suplementation

INTERVENTIONS:
Dietary Supplement: honey supplementation — honey supplementation
  Arms: honey group; malnourished control group

SUMMARY:
This study was a randomized single blinded case control prospective intervention study.

DETAILED DESCRIPTION:
Fifty infants and children of both sexes, aged 6 months to 3 years, with malnutrition were consecutively recruited from the Nutrition Clinic of the Pediatric Hospital, Ain Shams University.

These patients were randomly assigned following a simple randomization procedure (computerized random numbers) to either the honey group (group 1) or the malnourished control group (group 2) with a 1:1 allocation ratio. Each group consisted of 25 patients.

An additional 25 healthy infants and children with the same age range and of both sexes were recruited from the outpatient pediatric clinic of Ain Shams University, Egypt as a healthy control group (group 3).

The inclusion criteria was in whom the under nutrition is caused by inadequate energy intake, while the exclusion criteria included markedly ill patients, and children with chronic or severe systemic illness or malabsorption disorders, chromosomal aberrations, inborn errors of metabolism and cerebral palsy.

History taking with special emphasis on the dietetic history, history of any disease that might interfere with the nutrient intake or their use by the body and history of any acute or chronic illness. And full body Examination which include anthropometric measurements weight, height and mid arm circumference.

Each patient in the intervention group or honey group or group 1 took oral honey in a dose of 2ml/kg/day for 8 weeks; the calculated dose of honey was dissolved in water with a ratio of 1: 3, respectively, and then ingested by the patient before breakfast.

ELIGIBILITY:
Inclusion Criteria:

simple malnutrition

Exclusion Criteria:

cancer, sepsis, endocrine disorders, neurologic disorders, diabetes mellitus, heart failure renal failure liver cell failure. malabsorption disorders, chromosomal aberrations, inborn errors of metabolism cerebral palsy .

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
serum leptin | 2 month duration of honey supplementation
  effect of honey supplement on serum leptin in malnourished patients
anthropometric measurements | 2 month duration of honey supplementation
  effect of honey on growth assessed by anthropomerty

SECONDARY OUTCOMES:
frequency of infection and total caloric intake in the honey group | 2 month duration of honey supplementation
  compare effect of honey on frequency of infection in supplemented group compared to malnourished on rehabilitation